CLINICAL TRIAL: NCT05432063
Title: Evaluation of Reliability and Validity of Urdu Version of Oxford Shoulder Score Scale Among Pakistani Population
Brief Title: Urdu Version of Oxford Shoulder Score Scale: Reliability and Validity Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00261
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Shoulder Pain
Keywords: Oxford Shoulder Score Scale; Urdu Version; Reliability; Validity; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this study is to translate and culturally adapt the Oxford Shoulder Score Scale into Urdu, as well as to assess its reliability and validity in the Urdu-speaking Pakistani community. This research will also look at the relationship between Oxford Shoulder Score Scale and the Shoulder Pain And Disability Index and Short Form - 36 scores for shoulder pain.

DETAILED DESCRIPTION:
The English version of the Oxford Shoulder Score Scale will be translated and culturally modified into Urdu. The Oxford Shoulder Score Scale, as well as other correlation measures, will be disseminated among 104 individuals in the Pakistani Urdu speaking community, who will be chosen using a convenience sample approach and based on pre-defined inclusion and exclusion criteria. For the intra- and inter-observer validity and reliability of the Oxford Shoulder Score Scale, Shoulder Pain And Disability Index, and Short Form - 36, questionnaires will be filled on the same day by two observers, with a two-hour gap between the first and second application. This is the inter-observer evaluation. The third application for the intra-observer evaluation will be completed after 7 days. Statistical Package of Social Sciences Version 26 will be used to enter and analyses the data. The internal consistency will be assessed using the Cronbach alpha value. The test-retest reliability will be assessed using an inter-class correlation coefficient. The content validity, criteria and construct validity, as well as responsiveness, of the Oxford Shoulder Score Scale scale will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Documented cognitive impairment
* Patient with shoulder instability
* Acute traumatic shoulder injury

Exclusion Criteria:

* Age under 18 years
* Recent surgery
* Pain origination from neoplasms
* Systemic arthritic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pakistani general population with shoulder pain.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score Scale | 1st day
  The OSS is a 12-item questionnaire that patients with a degenerative or inflammatory shoulder disease must complete. Each question includes five response options, each with a score range from 0 to 4. The overall score runs from 0 to 48 (worst to greatest).
Shoulder Pain And Disability Index | 1st day
  The Shoulder Pain And Disability Index is a self-report questionnaire that evaluates pain and impairment in the shoulder. It is made up of 13 items divided into two subscales: pain (5 items) and disability (5 items) (8 items). Both subscales' items are rated on a scale of 0 to 10 (no pain or impairment) (the worst imaginable pain or so much difficulty on performing tasks that help is required).
Short Form - 36 | 1st day
  The SF-36 is a 36-question Health Related Quality of Life survey divided into eight sections: vitality, physical functioning, bodily pain, general health, physical role functioning, emotional role functioning, social role functioning, and mental health. Each component of the questionnaire can be given a score ranging from 0 to 100. The lower the score, the lower the quality of life for the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No